CLINICAL TRIAL: NCT04978688
Title: A Randomized Open Label Study to Evaluate the Safety, PK, and PD of Relugolix Alone and Relugolix Combined With Hormonal Add-Back Therapy for 6 Weeks in Healthy Premenopausal Female Subjects
Brief Title: Study of Relugolix Alone and Relugolix Combined With Hormonal Add-Back Therapy in Healthy Premenopausal Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Myovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MVT-601-1001
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
MeSH Terms: interventions — relugolix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Relugolix (Experimental): Participants received relugolix 40 milligrams (mg) alone for 6 weeks.
  Interventions: Drug: Relugolix
- Relugolix + E2/NETA (Experimental): Participants received relugolix 40 mg and E2/NETA at 1 mg/ 0.5 mg for 6 weeks.
  Interventions: Drug: Relugolix; Drug: E2/NETA

INTERVENTIONS:
Drug: Relugolix — Administered as an oral tablet once daily.
Drug: E2/NETA — Administered as an oral tablet once daily.
  Arms: Relugolix + E2/NETA

SUMMARY:
This was a randomized, open-label, repeat dose study of once daily relugolix alone or relugolix combined with hormonal add-back therapy (combination estradiol/norethindrone acetate) (E2/NETA) to assess safety, including markers of bone resorption, pharmacokinetics (PK), and pharmacodynamics (PD) endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal female between 18 and 48 years of age.
2. E2, P, LH and FSH concentrations within 0.5x of the lower limits of normal range and 2x of the upper limits of normal upper limits of normal range (ULN)
3. Regular menstrual periods for the 3 months prior to study enrollment
4. Body weight ≥ 45 killograms (kgs) and body mass index (BMI) of 20 to 36
5. Capable of giving written informed consent

Exclusion Criteria:

1. Pregnancy
2. Lactating Females
3. Any contraindication to the treatment with E2 and NETA
4. Use of the following medications in the 3 months prior to screening: injectable hormonal contraceptives, sex hormone medications or danazol
5. Use of the following medications in the 6 months prior to screening: injectable gonadotropin-releasing hormone agonists, hormonal, or non-hormonal intrauterine devices
6. History of sensitivity to any of the study medications of components thereof or history of drug
7. Significant gynecological, endocrine, metabolic or other health conditions
8. History of regular alcohol consumption within 6 months of study

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2016-09-21 (Actual); Study Completion 2016-09-21 (Actual)

PRIMARY OUTCOMES:
PK: Area Under The Concentration-Time Curve From Time Zero To Hour 24 (AUC0-24) Of Relugolix, E2, Estrone (El), Ethinylestradiol (EE), NETA | Predose and up to 24 hours at Weeks 3 and 6
PK: Maximum Concentration (Cmax) Of Relugolix, E2, El, NETA | Predose and up to 24 hours at Weeks 3 and 6
PK: Time To Maximum Concentration (Tmax) Of Relugolix, E2, El, EE, NETA | Predose and up to 24 hours at Weeks 3 and 6

SECONDARY OUTCOMES:
Change From Baseline In Serum Follicle Stimulating Hormone (FSH) At Week 6 | Baseline, Week 6
Change From Baseline In Serum Luteinizing Hormone (LH) At Week 6 | Baseline, Week 6
Change From Baseline In Serum Progesterone (P) At Week 6 | Baseline, Week 6
Change From Baseline In Serum E2 And E1 At Week 6 | Baseline, Week 6
Change From Baseline In N-telopeptide And C-telopepetide Concentrations At Week 6 | Baseline, Week 6
Incidence Of Treatment-Emergent Adverse Events | 8 weeks
Incidence Of Hot Flush | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Lukes A, Migoya E, Johnson B, Lee TY, Li Y, Arjona Ferreira JC. A Randomized Open-Label Study of Relugolix Alone or Relugolix Combination Therapy in Premenopausal Women. Clin Pharmacokinet. 2023 Aug;62(8):1169-1182. doi: 10.1007/s40262-023-01269-9. Epub 2023 Jun 26. PMID 37365436